CLINICAL TRIAL: NCT01161693
Title: The Effects of a Head Elevated Ramped Position During Elective Cesarean Delivery After Combined Spinal Epidural (CSE) Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Joanne Douglas, MD, FRCPC, University of British Columbia, Department of Anesthesia, BC Women's Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H10-01157
Record Dates: First submitted 2010-07-12; First posted 2010-07-13 (Estimated); Last update posted 2011-08-10 (Estimated); Status verified 2011-08

CONDITIONS: Cesarean Section
Keywords: Cesarean section; spinal anesthesia; CSE; ramped up position; TROOP pillow; elevation pillow; maternal comfort; Maternal Comfort after CSE during elective Cesarean Section in relation to adequate height of Anesthetic Block

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Standard pillow under head (No Intervention): Control (C) - Standard pillow under head (figure 1) as is the usual practice at BC Women's Hospital
  Interventions: Device: TROOP® elevation pillow
- Troop Elevation Pillow in horizontal position-HERP (Active Comparator): TROOP® elevation pillow (designed by an American bariatric anaesthesiologist Dr Craig Troop, plastic covered foam pillow with an elevation angle of 20 degrees which can simply be placed on the operating table)
  Interventions: Device: TROOP® elevation pillow
- Troop Elevation Pillow in horizontal position-HERP-H (Active Comparator): Operating table tilted in Trendelenberg position so angle of Troop pillow is parallel to floor (figure 3) until establishment of adequate block and then the bed levelled to horizontal i.e. to the same position as group (HERP) (figure 2)
  Interventions: Device: TROOP® elevation pillow

INTERVENTIONS:
Device: TROOP® elevation pillow — Maternal Comfort after CSE during elective Cesarean Section in relation to adequate height of Anesthetic Block
  Arms: Standard pillow under head
Device: TROOP® elevation pillow — designed by an American bariatric anaesthesiologist Dr Craig Troop, plastic covered foam pillow with an elevation angle of 20 degrees which can simply be placed on the operating table
  Arms: Troop Elevation Pillow in horizontal position-HERP
Device: TROOP® elevation pillow — designed by an American bariatric anaesthesiologist Dr Craig Troop, plastic covered foam pillow with an elevation angle of 20 degrees which can simply be placed on the operating table
  Arms: Troop Elevation Pillow in horizontal position-HERP-H

SUMMARY:
This study will randomly allocate 180 women undergoing elective C-sections under combined spinal epidural (CSE) Anesthesia at BC Women's Hospital to one of three groups: Standard Pillow under Head (Control), Head Elevated in Ramped Position immediately after regional anesthesia (HERP), or Head Elevated Ramped Position horizontally- Horizontal until establishment of anesthesia and then head elevated for the surgical procedure (HERP-H). The subjects will be monitored for blood pressure changes (hypotension), comfort levels and time to adequate level of the anesthetic block obtained with the CSE. The study will determine if positioning a parturient in the ramped position using an elevation pillow will significantly increase the time for anesthesia to reach the dermatome level of T4 as well as whether it increases maternal comfort and provides a better airway position for the parturient.

DETAILED DESCRIPTION:
The majority of elective and emergency cesarean deliveries are done under neuraxial anesthesia (spinal, epidural, combined spinal epidural) where the nerves to the lower half of the body are anesthetised with local anesthetic injected into the spine by the anesthesiologist. The injection is done at a low level in the spine and the local anesthetic rises within the cerebrospinal fluid to "block" or "freeze" higher nerves. The maximum level of sensory block anesthesia is determined by the cephalad distribution of the local anesthetic in the CSF, the total dose administered and uptake by neuronal tissue. The height of block is important to ensure that the woman is comfortable during cesarean delivery; generally a loss of cold sensation to ice at the dermatome level of T4 (the level of the nipples) is considered appropriate to commence surgery. If the block is below the level of T4, the woman is likely to feel discomfort and potentially pain, whereas too high a level can result in hemodynamic instability and difficulty breathing.

Conventionally patients are positioned on the operating table for surgery in a flat or horizontal (supine) position with a pillow under the head and a wedge positioned under the right hip to prevent aortocaval compression. Many women find lying completely flat while awake very uncomfortable and it is not uncommon for them to request that the head of the bed be elevated for comfort.

Difficult or failed intubation in obstetrics has been responsible for a number of maternal deaths over the years. The incidence of failed intubation is approximately 1 in 280 in the obstetric population compared to 1 in 2230 in the general surgical population. This is the result of a number of factors, including increased airway swelling due to progesterone. However, much of the perceived difficulty is due to anatomical factors such as increased breast size obstructing the levering hand when trying to insert the laryngoscope into the anesthetised patient's mouth. There have been numerous reports of similar problems with intubating the airway in bariatric (obese) parturients but recently the myth of obesity causing a difficult airway has been debunked providing the patient is positioned properly. Correct positioning of the patient in a "ramped" position with the patients head clearly elevated above their shoulders improves laryngeal exposure in obese patients. Collins et al. showed that "ramping" the patient until there was horizontal alignment between the external auditory meatus and sternal notch improved the laryngeal view when compared to the standard "sniff" position. Other benefits of the "ramped" position include better pre-oxygenation and bag mask ventilation in the 25 degree head up position than in the supine position in the severely obese patient. Studies in term parturients have shown an increase in the functional residual capacity (FRC) and slower desaturation rates in the head up position compared to the supine position. Some parturients require general anesthesia and endotracheal intubation for caesarean delivery. This may be due to the urgency of the situation, failure of neuraxial anesthesia or due to prolonged, difficult surgery. Having the woman adequately positioned for possible induction of general anesthesia, even though she is having a neuraxial technique, would be ideal and perhaps safer.

The ramped position can be achieved a number of ways including folded blankets stacked under the patient's body, neck and head. Most operating tables can be manipulated using the electronic or manual controls into a back/trunk up position. Commercial devices have been designed including the TROOP® elevation pillow, designed by an American bariatric anesthesiologist Dr Craig Troop. It is a plastic covered foam pillow with an elevation angle of 20 degrees which can simply be placed on the operating table. For the purposes of standardization we will be using the TROOP pillow as a means of achieving head elevation.

Taking these factors into consideration it would seem sensible to head elevate the parturient when positioned on the operating table. However, as the majority of obstetric surgeries are done under neuraxial anesthesia with only 1% undergoing general anesthesia in the elective situation and 3% in the emergency situation, the concern is that the position may result in a slower rise of the anesthetic block thereby delaying the start of surgery. The factors affecting the level of the anesthetic block are variable; gravity may play a part and the action of raising the head of parturient might logically result in a slower rise of anesthetic block resulting in an inadequate level for surgery, particularly with the commonly used hyperbaric local anesthetic. However, there is a large variability in patients and factors including dural sac compression from epidural venous plexus engorgement secondary to a degree of venal caval compression in the supine wedged position which may push the local anesthetic in a cephalad direction, and this may play a more significant role than simple gravity.

The effect of the ramped positioning on the level of spinal anesthesia has not been studied. Much of the work has been to look at the effects of lateral versus sitting posture for insertion of the spinal anesthetic on rise of block and hemodynamic stability. These studies showed a slower onset of anesthesia in the sitting group versus lateral with conflicting results in reduction in hypotension. The slower rise may be beneficial in preventing hemodynamic instability. Mardirosoff et al., when looking at the effects of sensory block extension during CSE in non obstetric patients, showed no significant change in block level when patients were sitting for 5 minutes following subarachnoid anesthesia; the mean level of block in all groups was to T4.

As there is no strong evidence either to support or oppose the rise of block against gravity, we will be doing a CSE anesthetic so that should the spinal block not rise to a sufficient level in any of the groups we will be able to supplement the block with local anesthetic injected into the epidural space to help raise the block by epidural volume expansion and/or by local anesthesia of the spinal nerves in the epidural space.

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy greater than 37 weeks gestation
* ASA (American Society of Anaesthesiologists) I and II classification of health. Class I a normal healthy patient and II a patient with mild systemic disease (i.e. mild asthma)
* Mothers presenting to the assessment unit with ruptured membranes or in the early stages of labour for whom a vaginal birth was not planned and who are therefore in need of urgent cesarean delivery.
* Potential subjects need to be able to read and understand English, unless an independent translator is available.

Exclusion Criteria:

* Women having general anesthesia
* Mothers in active labour - 3cm or more dilated with regular coordinated contractions (3 in 10 minutes)
* ASA classification 3 or above
* Emergency cesarean delivery for fetal heart rate abnormalities
* Maternal age <19
* BMI >40. Obesity makes it more difficult to site the combined spinal epidural which could lead to delay in positioning the patient quickly following subarachnoid block. Obesity can result in increased venal caval compression in the supine wedge position causing epidural venous plexus engorgement and dural sac compression which may result in a high block. A later study will look at the effects of positioning in the obese patient
* Mothers with a history of known tolerance to opioids
* Uterine over distension- polyhydramnios, twin pregnancy and estimated fetal weight of over 4kg by ultrasound scan -Uterine over distension can result in increased aortocaval compression which may lead to engorgement of the epidural venous plexus and dural sac compression which may result in a high block.
* Height over 180cm and below 150cm
* Women presenting for urgent caesarean delivery will be excluded if there is less than 60 minutes between the time that the researcher can approach them regarding the study and the time that they will have their surgery.

Min Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-07; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
length of time for anesthetic block to reach T4 | 11 months
  Our primary outcome is the length of time for anesthetic block to reach T4 from time of subarachnoid injection of local anesthetic, tested with ice

SECONDARY OUTCOMES:
Need for epidural supplementation | 11 months
  Need for epidural supplementation Maximum block height Maternal comfort Height of Block at 120 minutes Incidence of hypotension and dose of vasopressor used. Optimal head positioning for intubation - External Auditory Meatus/sternal relationship.

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Douglas, MD, FRCPC, Principal Investigator — University of British Columbia
Locations (1):
- BC Women's Hospital, Dept of Anesthesia, Vancouver, British Columbia, Canada